CLINICAL TRIAL: NCT00440245
Title: Bronchoprotection of Salbutamol in Asthma and COPD
Brief Title: Bronchoprotection of Salbutamol in Asthma and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bio-REB 06-231
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- salbutamol (Other): There are two groups, asthma and COPD, which are being compared with respect to bronchoprotection from an active treatment (salbutamol).
  Interventions: Drug: salbutamol

INTERVENTIONS:
Drug: salbutamol — 200 micrograms salbutamol from MDI

SUMMARY:
This study will investigate potential differences in how two puffs of salbutamol protects airway smooth muscle from contracting in people with asthma and chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
In asthma, the administration (inhalation) of a selective β2 receptor agonist (e.g. salbutamol), prior to methacholine challenge has been shown to shift the dose response curve to the right and "bronchoprotect" the airway against airway smooth muscle contraction. The extent of β2 receptor agonist bronchoprotection in COPD is unknown.

Airway hyperresponsiveness (AHR) to direct acting agents such as histamine and methacholine is a feature of both asthma and COPD. In asthma, the abnormality leading to AHR is believed to be due to changes in airway smooth muscle (e.g. hypertrophy, hyperplasia, contractile apparatus) whereas in COPD the AHR is likely due to structural or geometric changes.

The investigators hypothesize that the bronchoprotection afforded by salbutamol against methacholine challenge will be greater in asthma than in COPD due to differences in underlying airway abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* asthma or COPD

Exclusion Criteria:

* asthma and COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
methacholine PC20 dose shift | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Donald Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No